CLINICAL TRIAL: NCT02678078
Title: Characterization of Cancer Tissue Using 3D Biosynthetic Material
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Technion, Israel Institute of Technology (Other)
Collaborators: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Dror Seliktar, Professor, Technion, Israel Institute of Technology
Other Study IDs: 0671-15-RMB
Record Dates: First submitted 2016-02-04; First posted 2016-02-09 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-05

CONDITIONS: Cancer
Keywords: cancer; diagnosis; biopsy; chemotherapy drugs; tumor
MeSH Terms: conditions — Neoplasms; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — we will collect a liver biopsy and blood
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Analyzing biopsy samples — Analyzing biopsy samples that is preformed as part of the patient treatment.

SUMMARY:
Characterization of Cancer Tissue Using 3D Biosynthetic Materials. Using liver biopsy from stage 4 cancer patients, the investigators will evaluate and characterize the metastatic cells.

DETAILED DESCRIPTION:
The investigators' biomaterial lab has developed an in vitro diagnostic system in which a cancer tumor is placed inside a 3D hydrogel. This material has similar properties to the human tissue and can visualize cell migration and proliferation. In this system, the investigators have already characterised human metastatic cells obtained from nude mice tumors. The diagnostic assay is able to evaluate the reduction in cell growth associated with anti-cancer drug therapy. The next step is to test the in vitro diagnostic system using human tissue samples from human patients, and to validate the system as a simple and effective a priori diagnostic tool for characterizing patient tumours.

ELIGIBILITY:
Inclusion Criteria:

* liver tumor

Exclusion Criteria:

* refuse to volunteer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: every man or women 18 years old or older, with a liver tumor.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
cell growth | 1 week
  biopsy will be placed inside 3D gel, and growth will be measured over 1 week time.

CONTACTS AND LOCATIONS:
Overall Officials: Dror seliktar, Prof, Study Director — Technion, Israel Institute of Technology
Locations (1):
- Rambam, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Yes